CLINICAL TRIAL: NCT00429494
Title: Phase II Study of GnRH Analogue for Ovarian Function Preservation in Hematopoietic Stem Cell Transplantation Patients
Brief Title: GnRH Analogue for Ovarian Function Preservation in Hematopoietic Stem Cell Transplantation Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-710
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-05

CONDITIONS: Amenorrhea; Premature Ovarian Failure; Ovarian Function Insufficiency
Keywords: Hematopoietic Stem Cell Transplantation; GnRH Analogue; Gonadotropin-releasing hormone analogue; GnRH-a; Ovarian Function; Fertility; Leuprolide Acetate; Lupron Depot; premature ovarian failure; POF; Abnormal suppression of menstruation; absence of menstruation
MeSH Terms: conditions — Amenorrhea; Primary Ovarian Insufficiency | interventions — Leuprolide; Surveys and Questionnaires; Hematopoietic Stem Cell Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leuprolide Acetate (Experimental): Leuprolide Acetate 22.5 mg intramuscular (IM) injection 2 months before hematopoietic stem cell transplantation (HSCT) transplant and 3 months post-transplant.
  Interventions: Drug: Leuprolide Acetate; Behavioral: Questionnaire; Procedure: Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: Leuprolide Acetate — 22.5 mg IM injection 2 months before transplant and 3 months post-transplant.
  Other Names: Leuprolide Acetate (delayed release); Lupron Depot
Behavioral: Questionnaire — Questionnaires taking about 15 minutes to complete.
  Other Names: Survey
Procedure: Hematopoietic Stem Cell Transplantation — Stem cell infusion on Day 0.
  Other Names: HSCT; Stem Cell Transplant

SUMMARY:
Primary Objectives:

* To determine the effectiveness of the 3-month depot leuprolide in inducing and maintaining secondary amenorrhea in patients undergo hematopoietic stem cell transplantation.
* To determine the incidence of regained ovarian function manifested as spontaneous restoration of menstruation and normalization of hormonal level in patients after transplantation and discontinuation of long-acting leuprolide.

DETAILED DESCRIPTION:
All participants in this study will be scheduled for hematopoietic stem cell transplantation at The University of Texas (UT) MD Anderson Cancer Center.

Within two months before the transplantation, all participants will have a medical history, physical exam, and blood tests for ovarian function and platelet count. Participants will also need to have a gynecologic exam within one year before the transplantation.

Participants who are eligible will receive the first dose of leuprolide as an injection into either the shoulder muscle or the thigh muscle during their first clinic visit. Participants who have low platelet count will be given platelet transfusion before the injection.

Participants will then go on to have the transplantation as scheduled. Three months after the first dose of injection participants will have another clinic visit where blood tests for ovarian function will be performed. A second dose of the leuprolide will be given as an injection into the muscle at this visit. Again, if patients have low platelet count at that time, platelet transfusion will be given to patients before the injection. Participants will be given a checklist sheet for them to record any side effects while on the effect of leuprolide.

Three months after the last dose of the injection, patients will have the option to start taking or to resume oral contraceptive pills. Those who choose not to take or to resume oral contraceptive pills will be followed and observed for the return of menstrual or monthly cycles. Those who choose to take or to resume oral contraceptive pills, has to stop taking oral contraceptive pills for a period of 3-6 months starting 1 year after transplantation for us to assess the ovarian function.

During the period of follow up and observation of the return of menstruation, participants will be seen every two months either in the clinic or in the hospital if they are admitted. Participants will fill out questionnaires about their menstrual history at these visits. They should take about 15 minutes to complete. Blood tests for the ovarian function will also be done during these visits.

This is an investigational study. The drug used in this study is commercially available and has been approved by FDA for use in prostate cancer patients. Its use in this study is investigational. About seventy-five patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic stem cell transplantation candidate.
* Post-menarche female less than 40 years old.
* Premenopausal before the start of transplantation, or the start of oral contraceptive pills.
* Follicle-stimulating hormone (FSH) less than or equal to 20 IU/L and Luteinizing hormone (LH) less than or equal to 20 IU/L within 1 weeks of initiation of injection or the ovarian status is determined by Gynecology Oncology Service.
* Agree to stop any oral contraceptive pills for a period of 3-6 months starting 1 year post-transplant

Exclusion Criteria:

* Breast cancer
* Ovarian cancer
* Pregnancy
* Hypersensitivity to any Gonadotropin-releasing hormone (GnRH) analogs

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2002-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Cheng YC, Takagi M, Milbourne A, Champlin RE, Ueno NT. Phase II study of gonadotropin-releasing hormone analog for ovarian function preservation in hematopoietic stem cell transplantation patients. Oncologist. 2012;17(2):233-8. doi: 10.1634/theoncologist.2011-0205. Epub 2012 Jan 26. PMID 22282904
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 18, 2002 to November 21, 2008. All participants were recruited in medical clinics.
Pre-assignment Details: Of the 60 participants enrolled, one participant was excluded prior to treatment due to ineligibility.
Period: Overall Study
Arm/Group | Leuprolide Acetate
Started | 59
Completed | 44
Not Completed | 15
Not completed — Withdrawal by Subject | 9
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Groups:
- Leuprolide Acetate: Leuprolide Acetate 22.5 mg intramuscular (IM) injection 2 months before HSCT transplant and 3 months post-transplant.
Arm/Group | Leuprolide Acetate
Number analyzed (Participants) | 59
Age Continuous [Median (Full Range); unit: years] | 25 [17 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Secondary Amenorrhea Following 3-month Depot Leuprolide
Description: Hormonal profile blood tests including follicle-stimulating hormone (FSH) test, luteinizing hormone (LH) and estradiol levels done every two months with menstruation questionnaire, starting three months after the injection of the second dose of leuprolide until the restoration of spontaneous menstruation or the presence of ovarian failure. Any unexpected vaginal bleeding or side effects during the period covered by leuprolide injection, which is 6 months, is recorded by participants in a monitoring checklist sheet given to them.
Time Frame: 6 months
Population: Of the 59 patients who underwent HSCT, nine patients refused the second dose of leuprolide and were subsequently taken off study. Six patients died of either disease progression or transplantation-related complications before their ovarian function status was evaluated.
Measure: Number; unit: participants
Arm/Group | Leuprolide Acetate
Number analyzed (Participants) | 44
participants | 37

ADVERSE EVENTS:
Time Frame: 5 years and 6 months
Arm/Group | Leuprolide Acetate
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 9/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate (N=59)
Menopausal side effects (Reproductive system and breast disorders) | 9 — Menopausal side effects, including hot flushing, vaginal dryness, and mood swings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No